CLINICAL TRIAL: NCT01713543
Title: Multifactorial, Evidence-based Program of Screening, Risk Modification and Physical Therapy to Prevent Falls Among Vulnerable Elderly Recently Discharged From Hospital to the Community.
Brief Title: Community-based Falls Prevention Program for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government); Duke-NUS Graduate Medical School (Other); Singapore General Hospital (Other); Changi General Hospital (Other); Health Promotion Board, Singapore (Other Government); Agency for Integrated Care, Singapore (Other); Jurong Health Services (Unknown)
Responsible Party: Principal Investigator, Dr. David Matchar, Professor and Director, Program in Health Services & Systems Research, Duke-NUS, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSRG10MAY002
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Accidental Falls
Keywords: falls
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The intervention consists of a tailored physical therapy focused on progressive strength, balance and gait training for a period of 3 months.
  Interventions: Other: physical therapy
- Control Group (No Intervention): Usual care by physician.

INTERVENTIONS:
Other: physical therapy — Tailored physical therapy sessions to modify impairments in balance and/or gait and to transition high-risk participants to an evidence-based group exercise program.
  Other Names: Falls Prevention
  Arms: Intervention Group

SUMMARY:
Background: Falls are the leading cause of injury among older adults in Singapore, but falls among the elderly can be preventable and the risks are predictable. Translating this understanding of falls etiology into an integrated clinical and public health program that is accessible to the elderly is a critical health services delivery challenge.

Hypothesis: An evidence-based program of screening, risk modification and physical therapy delivered in a community setting will reduce recurrent falls incidence among a high-risk group of elderly recently discharged to the community.

Methodology: This randomized controlled trial targets patients seen at Emergency Department (ED) for a fall or fall-related injuries who are at least 65 years old and will be discharged to home. Upon signing the informed consent form, the participants will be followed up for nine months from the baseline assessment during which the participants are randomized into either a control or the intervention group. The participants in the intervention group will be provided with a multifactorial program of screening, risk modification and physical therapy focused on progressive strength, balance, and gait training either as an individualized program or a group setting in the community for the first three months from the date of randomization. The number of recurrent falls will be monitored via a falls prevention diary maintained by (or for) each participant.

DETAILED DESCRIPTION:
Objective:

To develop and demonstrate the feasibility and effectiveness of a multifactorial, community-based falls prevention program of screening, risk modification, and progressive physical therapy that targets vulnerable elderly Singaporeans at high-risk of falls.

Methodology:

This two-year, multi-center, two-arm, parallel group, randomized controlled trial will be divided into three phases: (1) pre-study, (2) intervention, and (3) analysis.

During the pre-study phase, overseas experts will train local physiotherapists and community health workers on how to administer and deliver the falls prevention program. Engaging hospital-based physiotherapists to deliver the home-based assessments and exercise programs will maximize the likelihood of long-term sustainability of the intervention program. In addition, manuals will be developed for physiotherapists to guide the evaluation risk factor assessments, home environment assessments, appropriate referrals to different health care providers, and selection of exercise programs that will be progressive, challenging and of optimal intensity and durations. Manuals for risk factor assessments will be shared with the blinded assessors.

The intervention phase will be divided into two phases: a three-month "Active Intervention Phase" and a six-month "Maintenance Phase." In the beginning of the active intervention phase, the participants in the intervention group will receive a detailed falls risk assessment at the baseline assessment by a physiotherapist. The risk factors that will be assessed are the following:

1. Poor vision: Referral to ophthalmologist for correction
2. Polypharmacy: Referral to AIC for management of medications if use of five or more medications
3. Environmental Hazards: Caregiver education and suitable recommendations according to the CDC guidelines to modify risk such as removal of rugs, change to safer footwear, use of non-slip bath mats, additional lighting at night.
4. Deficiencies in gait, balance or mobility: Physiotherapist-supervised program of gait training, balance and strengthening exercises In the analysis phase, the collected data will be analyzed. The primary outcome measure of the study is the number of fallers over the entire study period. The number of falls will be captured by a falls prevention diary maintained by (or for) each participant.

Procedures:

The elderly seen at ED for a fall or fall-related injury will be screened for participation of the study. Once the consent is taken, all study participants will be given an assessment by a physiotherapist at baseline which assesses sociodemographic characteristics, functional status measured by the Short Physical Performance Battery (SPPB), two-minute walk test, history of falls, cognitive impairment measured by the Montreal Cognitive Assessment (MoCA), quality of life (EQ-5D-5L and EQ-VAS), health care utilization, and medical history (polypharmacy, orthostatic vital signs, and self-reporting eyesight and hearing).

At the end of baseline assessment, the participants will be assigned either a control or the intervention group. Before the start of the exercise sessions, the participants in the intervention group will. Need to complete Physical Activity Readiness Questionnaire (PAR-Q) and a medical evaluation by a physician to ensure that the participants are fit for physical activity. Based on the SPPB score at baseline assessment, participants will be categorized as either high-risk (SPPB<6) or low-to-moderate-risk (SPPB>6) for falls. High-risk patients will be given an individualized PT-supervised program of physical therapy that specifically targets impairments that interfere with engaging in exercise in group setting. The goal of the tailored physical therapy sessions is to modify impairments and transition these patients to an evidence-based exercise program. Low-to-moderate-risk patients will be directly enrolled into an evidence-based group exercise program. The group exercise programs will be offered as one-hour sessions, twice weekly over the intervention period. At the end of the active intervention phase, these participants will transition to a maintenance phase in which they will be encouraged to continue with the exercise on their own and will also be referred to the Health Promotion Board's STEP program.

The participants will be asked at the end of the active intervention phase (three months from the date of randomization) and at the end of the study period (nine months from the date of randomization) about their functional status, history of falls, cognitive impairment, quality of life, health care utilization, and medical history by the blinded assessors. Recurrent falls incidence will be monitored by participants' self-reporting monthly falls diary as well as monthly phone calls conducted by the study coordinator during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Seen in the Emergency Department for a fall or injury related to a fall
* Able to follow 3 step commands
* Singapore citizen or Permanent Resident
* Living at home upon discharge
* Provision of informed consent
* If admitted to the hospital, the illness or disability is one from which they are expected to recover basic ADLs or weight bearing of the lower extremity within the next month

Exclusion Criteria:

* Those patients with severe physical and/or mental impairments which preclude participation in a program of physical therapy (as determined by a primary physician) will NOT be eligible for participation.
* Unable to participate in the exercise program due to conflicting schedules (e.g. full-time employment, on dialysis)
* Serious life limiting illness
* Patients seen at ED due to road traffic accidents
* Unable to walk even with assistance
* Not community dwelling prior to ED visit
* Total blindness
* Needs emergency inpatient surgery and, if admitted to the hospital, the illness or disability is one from which they are not expected to recover basic ADLs or weight bearing in the lower extremity within the next one month.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 354 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The number of fallers who have fallen at least once during the 9-month study period | 9 months

SECONDARY OUTCOMES:
The number of injurious falls and healthcare utilization | 9 months
  Injurious falls are the falls that resulted in participants' seeking medical attention or restricting their daily activities for at least 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: David B Matchar, MD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore

REFERENCES:
- [Background] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK; LEAPS Investigative Team. Protocol for the Locomotor Experience Applied Post-stroke (LEAPS) trial: a randomized controlled trial. BMC Neurol. 2007 Nov 8;7:39. doi: 10.1186/1471-2377-7-39. PMID 17996052
- [Derived] Matchar DB, Eom K, Duncan PW, Lee M, Sim R, Sivapragasam NR, Lien CT, Ong MEH. A Cost-Effectiveness Analysis of a Randomized Control Trial of a Tailored, Multifactorial Program to Prevent Falls Among the Community-Dwelling Elderly. Arch Phys Med Rehabil. 2019 Jan;100(1):1-8. doi: 10.1016/j.apmr.2018.07.434. Epub 2018 Aug 27. PMID 30165053
- [Derived] Pua YH, Ong PH, Clark RA, Matcher DB, Lim EC. Falls efficacy, postural balance, and risk for falls in older adults with falls-related emergency department visits: prospective cohort study. BMC Geriatr. 2017 Dec 21;17(1):291. doi: 10.1186/s12877-017-0682-2. PMID 29268720
- [Derived] Matchar DB, Duncan PW, Lien CT, Ong MEH, Lee M, Gao F, Sim R, Eom K. Randomized Controlled Trial of Screening, Risk Modification, and Physical Therapy to Prevent Falls Among the Elderly Recently Discharged From the Emergency Department to the Community: The Steps to Avoid Falls in the Elderly Study. Arch Phys Med Rehabil. 2017 Jun;98(6):1086-1096. doi: 10.1016/j.apmr.2017.01.014. Epub 2017 Feb 12. PMID 28202383